CLINICAL TRIAL: NCT02311946
Title: A Phase 1, Open-Label Fixed-Sequence 2-Period Crossover Study Of Palbociclib (pd-0332991) In Healthy Volunteers To Estimate The Effect Of Antacid Treatment On The Bioavailability Of A 125 Mg Single Dose Of Six Experimental Formulations Of Palbociclib Relative To Palbociclib Administration Alone Under Fasted Conditions
Brief Title: A Pilot Study To Investigate The Effect Of Concurrent Antacid Administration On The Bioavailability Of Six Experimental Formulations Of Palbociclib
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: A5481041
Record Dates: First submitted 2014-12-04; First posted 2014-12-09 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Healthy
Keywords: Palbociclib, Rabeprazole, Proton Pump Inhibitor, Drug Interaction Study, DDI
MeSH Terms: interventions — palbociclib; Rabeprazole; Proton Pump Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Cohort 1 (Experimental): Cohort 1 will receive a 125 mg round yellow palbociclib tablet containing succinic acid
  Interventions: Drug: Palbociclib Alone; Drug: Palbociclib + Rabeprazole
- Cohort 2 (Experimental): Cohort 2 will receive a 125 mg oval yellow palbociclib spray-dried dispersion tablet containing HMPC E3
  Interventions: Drug: Palbociclib Alone; Drug: Palbociclib + Rabeprazole
- Cohort 3 (Experimental): Cohort 3 will receive a 125 mg oval yellow palbociclib spray-dried dispersion tablet with HMPC E3 and succinic acid.
  Interventions: Drug: Palbociclib Alone; Drug: Palbociclib + Rabeprazole
- Cohort 4 (Experimental): Cohort 4 will receive a 125 mg oval white/yellow palbociclib bilayer tablet with tartaric and succinic acid.
  Interventions: Drug: Palbociclib Alone; Drug: Palbociclib + Rabeprazole
- Cohort 5 (Experimental): Cohort 5 will receive a 125 mg oval yellow palbociclib fluid bed granulation tablet with succinic acid.
  Interventions: Drug: Palbociclib Alone; Drug: Palbociclib + Rabeprazole
- Cohort 6 (Experimental): Cohort 6 will receive a 125 mg palbociclib oral solution
  Interventions: Drug: Palbociclib Alone; Drug: Palbociclib + Rabeprazole

INTERVENTIONS:
Drug: Palbociclib Alone — In Period 1 of each Cohort, a single 125 mg dose of palbociclib will be administered alone in a fasted state, and subjects will undergo serial pharmacokinetic blood sampling for up to 120 hours post-dose.
  Other Names: Palbociclib, PD-0332991
Drug: Palbociclib + Rabeprazole — In Period 2 of each Cohort, subjects will receive daily 40 mg oral doses of the proton pump inhibitor rabeprazole on 7 consecutive days. Approximately 4 hours after the last rabeprazole dose a single 125 mg dose of palbociclib will be administered alone in a fasted state, and subjects will undergo serial pharmacokinetic blood sampling for up to 120 hours post-dose.
  Other Names: Palbociclib, PD-0332991, Rabeprazole, Aciphex, Proton Pump Inhibitor, PPI

SUMMARY:
This study will investigate whether concurrent administration of rabeprazole, an antacid known as a proton pump inhibitor, alters the absorption of the drug palbociclib when given as one of six experimental formulations.

DETAILED DESCRIPTION:
This will be a 6 cohort study investigating one experimental formulation of palbociclib in each of the six cohorts of 10 healthy subjects. Each cohort will receive two treatments in a fixed-sequence. In Period 1, all subjects will receive a single 125mg dose of palbociclib alone and undergo serial pharmacokinetic blood sampling for up to 120 hours post-dose. In Period 2, all subjects will receive daily 40mg doses of Rabeprazole for 7 consecutive days, and approximately 4 hours after the Day 7 rabeprazole dose each subject will receive a single 125mg dose of palbociclib. Subjects will undergo serial pharmacokinetic blood sampling up to 120 hours post-dose.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Male or Female of non-childbearing potential,
* Having a body weight >50 kg
* Having a bopy mass index (BMI) between 17.5 and 30.5 kg/m2.

Exclusion Criteria:

* Any condition possibly affecting drug absorption (eg, gastrectomy)
* A positive urine drug or cotinine test
* A known history of hypersensitivity to palbociclib
* A supine systolic blood pressure >140 mmHg, or a QTc >450 msec.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2015-01; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
AUCinf | Pre-dose to 120 hours post-dose
  Area under the concentration-time curve from time zero to infinity.
Cmax | Pre-dose to 120 hours post-dose
  Maximum observed plasma concentration

SECONDARY OUTCOMES:
AUClast | Pre-dose to 120 hours post-dose
  Area under the concentration-time curve from time zero to the time of the last quantifiable concentration.
CL/F | Pre-dose to 120 hours post-dose
  Apparent oral clearance from plasma
Tmax | Pre-dose to 120 hours post-dose
  Time of the maximum observed concentration post-dose.
Vz/F | Pre-dose to 120 hours post-dose
  Apparent volume of distribution
t1/2 | Pre-dose to 120 hours post-dose
  Terminal phase half-life

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (3):
- United States (3):
  - MRA Clinical Research - Phase 1, Miami, Florida
  - Miami Research Associates, LLC, South Miami, Florida
  - MRA Clinical Research, LLC, South Miami, Florida